CLINICAL TRIAL: NCT07054112
Title: Efficacy of Live Online Course Mindfulness Program on Perceived Fatigue in Hemodialysis Patients
Acronym: MEDIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR240292
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: chronic kidney desease; MBSR program; fatigue; Song scale
MeSH Terms: conditions — Fatigue | interventions — Mindfulness-Based Stress Reduction; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients receive an MBSR (Mindfulness on Stress Reduction) meditation program delivered by a certified instructor.
  Interventions: Other: Mindfulness-Based Stress Reduction (MBSR) meditation program
- Control group (Other): Patients will be in a wait list group. They will receive their usual care during the study follow-up. Between M8 and M10 they will receive a MBSR meditation program
  Interventions: Other: Control group

INTERVENTIONS:
Other: Mindfulness-Based Stress Reduction (MBSR) meditation program — The sessions of the meditation program (Mindfulness on Stress Reduction) will be delivered online, outside of the dialysis sessions. They will receive standard care during their hemodialysis sessions.
  The program is composed of 8 sessions of 2h30 + 1 day of mindfulness, during 2 months.
  Arms: Experimental group
Other: Control group — Patients in the control group will be in a wait list group. They will receive standard care during their hemodialysis sessions. they will receive the MBSR meditation program between M8 and M10.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to assess the efficacy of a 2-month live online mindfulness meditation program in reducing perceived fatigue (measured by the SONG-HD Fatigue Scale) in patients undergoing chronic hemodialysis.

The sponsor expects that a live online mindfulness meditation course will have a significant public health impact by reducing perceived fatigue, which is strongly associated with cardiovascular events, mortality, and reduced quality of life.

Participants will be enrolled according to eligibility criteria and randomized into one of the following groups:

Experimental group: will receive an 8-week live online Mindfulness-Based Stress Reduction (MBSR) program.

Control group: will receive standard care during their hemodialysis sessions and will be offered the same live online MBSR program between months 8 and 10.

Patients will complete self-administered questionnaires at baseline, 2 months, 8 months, and 10 months to monitor changes in fatigue, anxiety, and quality of life.

DETAILED DESCRIPTION:
Chronic kidney disease requiring a replacement therapy is a main public health issue. The overall incidence of treated end-stage renal disease is 169 per million inhabitants in France (Annual REIN report, Biomedicine Agency, 2021). Chronic kidney disease patients requiring a replacement therapy have a very increased mortality compared to the general population and their quality of life is particularly impacted.

The international initiative Standardized Outcomes in Nephrology hemodialysis (SONG-HD) has identified and prioritized the most important outcomes for patients requiring hemodialysis. The patients, their caregivers and health professionals have highlighted that perceived fatigue is one of the biggest issues once the hemodialysis began. Fatigue is a complex and subjective experience which include physical (muscular weakness, low stamina) and psychological symptoms (feeling of increased effort and decrease cognitive endurance). For patients with chronic hemodialysis, additionally to the burden of disease, they must receive in average three dialysis sessions per week which is a source of exhaustion. Fatigue is associated with an increase of cardiovascular events, an increase of mortality, a reduction of quality of life and consequently a less good compliance to dialysis. The outcome "fatigue" is then one of the critically important outcomes which must be assessed in all clinical trials and the investigators need to explore interventions to improve well-being of patients and to prevent patient's exhaustion.

Mindfulness meditation is defined as moment to moment self-regulation of attention. This practice helps cultivate non-judgmental acceptance of the present moment. Besides, a cognitive behavioral therapy including meditation significantly improve the well-being, the mood, the anxiety and stress perception of chronic hemodialysis patients. Several studies have showed that mindfulness meditation is associated with a decrease of systolic blood pressure, a decrease of depressive symptoms and an increase in self-compassion scores in hemodialysis patients.

Numerous studies have shown a significant improvement in fatigue thanks to a mindfulness meditation program in patients with lung cancer, breast cancer, in healthcare workers facing fatigue linked to empathic distress or even in volleyball athletes presenting moral fatigue linked to strong competition. However, to our knowledge, there is no study assessing the impact of a mindfulness meditation program on fatigue patients receiving chronic hemodialysis.

The investigators hypothesize that mindfulness meditation could regulate the psychological and physical perceived fatigue of hemodialysis patients. Meditation provides techniques allowing the participant to learn to step back from emotions, thoughts and experience in general. This is the decentring process. Furthermore, yoga, which is a part of the program, can help regulate the physical aspects of fatigue by leading to an increase in muscle mass and cardiac activity.

Benefit/ risk balance Non-invasive test. Very favorable benefit/risk balance, taking into account the demonstrated benefits in terms of stress and fatigue management of mindfulness meditation programs.

Absence of serious adverse effects reported under normal conditions while respecting the usual contraindications corresponding to the inclusion criteria.

A recent research showed that practicing mindfulness meditation is associated with transient distress and negative impacts at rates similar to other psychological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Written informed consent obtained from the participant
* Patients on chronic hemodialysis for more than 3 months
* Participant affiliated to social security system
* Internet access
* Patient motivation/commitment
* Patient having 3 days of dialysis per week

Exclusion Criteria:

* Major acute depression
* Patient on peritoneal dialysis
* Already participated in an MBSR program
* Patients covered by articles L1121-5 to L1121-8 of the French Public Health Code (corresponding to protected persons: pregnant women, women who have recently given birth or are breastfeeding, persons deprived of their rights by judicial or administrative decision, minors, and persons benefiting from legal protection: curatorship or guardianship).
* Planned hospitalization within 4 months
* Known cognitive disorder (Mini Mental State Evaluation <23 for more than 65 years)
* Known schizophrenia
* Known psychotic personality disorder
* Suicide attempt or suicidal ideation
* Addiction to alcohol or drugs during addiction treatment
* Cancer undergoing chemotherapy
* Pathological grieving process
* Compulsive eating disorders
* No understanding of French
* Unaided deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in the SONG-HD fatigue scale between baseline and 2 months follow-up. | Between baseline and 2 months follow-up.
  SONG-HD scale means Standardised Outcomes in Nephrology-Haemodialysis; The score will vary from 0 to a maximum of 9

SECONDARY OUTCOMES:
Evolution of the score on the SONG-Fatigue scale between baseline, M2, M8 and M10 | between baseline, Month-2, Month-8 and Month-10
  SONG-HD scale means Standardised Outcomes in Nephrology-Haemodialysis; The score will vary from 0 to a maximum of 9
Evolution of MFI score between baseline, M2, M8 | between baseline, Month-2, Month-8
  MFI means Multidimensional Fatigue Inventory. The score will vary from 0 to a maximum of 100
Evolution of quality of life (KDQOL) at baseline, M2, M8 | at baseline, Month-2, Month-8
  KDQOL means Kidney Disease Quality of Life
Evolution of anxiety (HAD) between baseline, M2, M8 | between baseline, Month-2, Month-8
  HAD means Hospital Anxiety and Depression scale. The HAD scale is a screening instrument for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21).
Evolution of Mindfulness Score (FFMQ) between baseline, M2 and M8 | between baseline, Month-2 and Month-8
  FFMQ means Five Facet Mindfulness Questionnaire. It comprises 39 questions. Each item ranges from 1 to 5.
The occurrence of cardiovascular events at M8 | at Month-8
Mortality at M8 | At Month-8
The number of vascular access events at M8 | At Month-8

CONTACTS AND LOCATIONS:
Overall Officials: Marine NAUDIN, PhD, Principal Investigator — CHRU de Tours
Locations (10):
- France (10):
  - CH Angers, Angers
  - CH Bayonne, Bayonne
  - CHRU de Bordeaux, Bordeaux
  - AIRBP 28, Chartres
  - AURAD Aquitaine, Gradignan
  - CHD Vendée, La Roche-sur-Yon
  - ECHO Nantes, Nantes
  - ATTIRO Orléans, Orléans
  - CHRU De Tours, Tours
  - CALYDIAL, Vienne

IPD SHARING:
Plan to Share IPD: No